CLINICAL TRIAL: NCT04640532
Title: An Open-Label, Multicenter, Phase 1b/2 Study of the Safety and Efficacy of KRT-232 in Combination With TL-895 for the Treatment of Relapsed or Refractory Myelofibrosis and KRT-232 for the Treatment of JAK Inhibitor Intolerant Myelofibrosis.
Brief Title: KRT-232 in Combination With TL-895 for the Treatment of R/R MF and KRT-232 for the Treatment of JAKi Intolerant MF
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kartos Therapeutics, Inc. (Industry)
Collaborators: Telios Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KRT-232-113
Record Dates: First submitted 2020-11-17; First posted 2020-11-23 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Myelofibrosis; Post-PV MF; Post-ET Myelofibrosis; Primary Myelofibrosis
Keywords: Relapsed/Refractory Myelofibrosis; Janus associated Kinase Inhibitor-Intolerant Myelofibrosis; MDM2; navtemadlin
MeSH Terms: conditions — Primary Myelofibrosis | interventions — navtemadlin; 2-((3R,5R,6S)-5-(3-chlorophenyl)-6-(4-chlorophenyl)-1-((S)-1-(isopropylsulfonyl)-3-methylbutan-2-yl)-3-methyl-2-oxopiperidin-3-yl)acetic acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1 (R/R MF), Dose Level 1 (Experimental): TL-895 at 200 mg once a day (QD) continuously starting on Cycle 1 Day 1 in a 28-day cycle.
  KRT-232 240mg will be administered orally, once daily (QD), on days 1-7 in a 28-day cycle starting on Cycle 2 Day 1.
  Interventions: Drug: KRT-232; Drug: TL-895
- Cohort 1 (R/R MF), Dose Level 2 (Experimental): TL-895 at 300 mg once a day (QD) continuously starting on Cycle 1 Day 1 in a 28-day cycle.
  KRT-232 at 240mg will be administered orally, once daily (QD), on days 1-7 in a 28-day cycle starting on Cycle 2 Day 1.
  Interventions: Drug: KRT-232; Drug: TL-895
- Cohort 2 (R/R MF), Dose Level 1 (Experimental): TL-895 at 100 mg twice a day (BID) continuously starting on Cycle 1 Day 1 in a 28-day cycle.
  KRT-232 at 240mg will be administered orally, once daily (QD), on days 1-7 in a 28-day cycle starting on Cycle 2 Day 1.
  Interventions: Drug: KRT-232; Drug: TL-895
- Cohort 2 (R/R MF), Dose Level 2 (Experimental): TL-895 at 150 mg twice a day (BID) continuously starting on Cycle 1 Day 1 in a 28-day cycle.
  KRT-232 at 240mg will be administered orally, once daily (QD), on days 1-7 in a 28-day cycle starting on Cycle 2 Day 1.
  Interventions: Drug: KRT-232; Drug: TL-895
- Cohort 3 (JAKi Intolerant MF) (Experimental): KRT-232 at 240mg will be administered orally, once daily (QD), on days 1-7 in a 28-day cycle.
  Interventions: Drug: KRT-232

INTERVENTIONS:
Drug: KRT-232 — KRT-232, administered by mouth
Drug: TL-895 — TL-895, administered by mouth
  Arms: Cohort 1 (R/R MF), Dose Level 1; Cohort 1 (R/R MF), Dose Level 2; Cohort 2 (R/R MF), Dose Level 1; Cohort 2 (R/R MF), Dose Level 2

SUMMARY:
This study evaluates KRT-232 in Combination With TL-895 for the Treatment of Relapsed or Refractory Myelofibrosis and KRT-232 for the Treatment of JAK Inhibitor Intolerant Myelofibrosis.

DETAILED DESCRIPTION:
Cohorts 1 and 2 will undergo dose finding and dose expansion. Eligible patients will be randomly assigned to an open cohort, either Cohort 1 or Cohort 2. Cohort 3 will be conducted as a dose expansion, independent of Cohorts 1 and 2.

Cohort 1 will follow a 3+3 dose escalation design to determine the maximum tolerated dose (MTD)/maximum administered dose (MAD) and recommended Phase 2 dose (RP2D) of TL-895 administered QD in combination with KRT-232. A Safety Review Committee (SRC) will review the safety data during the dose escalation to decide on dose escalation and/or exploration of intermediate doses.

Cohort 2 will follow a 3+3 dose escalation design to determine the MTD/MAD and recommended RP2D of TL-895 administered BID in combination with KRT-232. An SRC will review the safety data during the dose escalation to decide on dose escalation and/or exploration of intermediate doses.

Cohort 3 will be conducted a 2-stage design. In stage 1, enrollment will continue until 15 evaluable patients have been enrolled. An SRC will review the data during the study and if there are ≥4 responders based on the futility criteria and safety data from Stage 1, Cohort 3 expansion will commence. If there are ≤3 patients responding to therapy, Cohort 3 will be terminated. Once expansion criteria have been met, Cohort 3 will be expanded to a total of 46 evaluable patients for Stage 2 analyses.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of primary MF, post-PV MF, or post-ET MF, (WHO 2016)
* ECOG ≤ 2
* Cohort 1 and Cohort 2: R/R following JAK inhibitor treatment
* Cohort 3: patients who are intolerant to JAK inhibitor treatment

Exclusion Criteria:

* Prior treatment with MDM2 inhibitors or p53-directed therapies
* Prior treatment with a BCR-ABL, phosphoinositide 3-kinase (PI3k), mammalian target of rapamycin (mTOR), bromodomain and extraterminal domain (BET), histone deacetylase (HDAC), or spleen tyrosine kinase (Syk) inhibitor
* Prior splenectomy
* Splenic irradiation within 3 months prior to the first dose of study treatment
* Clinically significant thrombosis within 3 months of screening
* Grade 2 or higher QTc prolongation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2020-11-17 (Actual); Primary Completion 2022-05-11 (Estimated); Study Completion 2025-07-24 (Estimated)

PRIMARY OUTCOMES:
Phase 1b - The MTD/MAD and RP2D of TL-895 in combination with KRT-232 in patients with R/R MF (Cohort 1 and Cohort 2) | 56 Days
  DLTs will be used to establish the MTD. RP2D will be determined by the SRC based on safety data from the combination of TL-895 and KRT-232.
Phase 2 - Spleen response rate for each cohort | 24 Weeks
  A reduction in spleen volume as assessed by MRI (or CT) ≥ 35% from baseline at Week 24

SECONDARY OUTCOMES:
Total Symptom Score (TSS) | 24 Weeks
  The change in TSS based Myelofibrosis Symptom Assessment Form version 4.0 (MFSAF v4.0)

CONTACTS AND LOCATIONS:
Locations (37):
- United States (6):
  - University of Alabama at Birmingham School of Medicine, Division of Hematology and Oncology, Birmingham, Alabama
  - The Oncology Institute of Hope, Whittier, California
  - Lake City Cancer Center, Lake City, Florida
  - Carle Cancer Center, Urbana, Illinois
  - Columbia University Medical Center, Fort Lee, New Jersey
  - Memorial Sloan Kettering Cancer Center (MSKCC), New York, New York
- Austria (2):
  - LKH Hochsteiermark, Leoben
  - Meduni Wien, Univ. Klinik für Innere Medizin I, Vienna
- Bulgaria (3):
  - University Multiprofile Hospital for Active Treatment Dr. Georgi Stranski, Pleven, Pleven
  - University Multiprofile Hospital for Active Treatment Dr. Georgi Plovdiv, Plovdiv
  - Hematology Clinic Specialized Hospital for Active Treatment of Hematological Diseases, Sofia, Sofia
- France (6):
  - Chu Amiens Picardie Site Sud, Amiens
  - CHU de Limoges Service Hématologie Clinique et Thérapie Cellulaire, Limoges
  - CHU Nantes - Hôtel Dieu, Nantes
  - CHU de Nice Hospital, Nice
  - Hôpital Saint Louis, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
- Germany (2):
  - University Hospital Halle (Saale), Department of Internal Medicine IV - Hematology and Oncology, Halle
  - University Hospital Marburg, Department of Hematology, Oncology and Immunology, Marburg
- Hungary (4):
  - Moritz Kaposi General Hospital, Department of Hematology, Kaposvár
  - Szabolcs-Szatmar-Bereg County Hospitals and University Teaching Hospital, Department of Hematology, Nyíregyháza
  - Medical Center of the University of Pecs, 1st Department of Internal Medicine, Division of Hematology, Pécs
  - Fejer County St. Gyorgy University Teaching Hospital, Department of Internal Medicine III, Hematology, Székesfehérvár
- Italy (5):
  - Polyclinic S. Orsola-Malpighi, Bologna
  - ASST Spedali Civili di Brescia, Brescia
  - Careggi University Hospital, Florence
  - Hospital Casa Sollievo della Sofferenza, Department of Oncology and Hematology, Division of Hematology, Foggia
  - Hospital of Ravenna, Operative Unit of Hematology, Ravenna
- Poland (5):
  - Jan Biziel University Hospital #2 in Bydgoszcz, Department of Hematology, Bydgoszcz
  - Pratia Onkologia Katowice, Katowice
  - Frederic Chopin Provincial Teaching Hospital No. 1 in Rzeszow, Department of Hematology, Rzeszów
  - Slupsk Provincial Specialist Hospital n.a. Janusz Korczak, Department of Hematology, Słupsk
  - Nasz Lekarz Medical Outpatient Clinics Slawomir Jeka, Torun
- Serbia (2):
  - Clinical Center of Serbia, Belgrade
  - Clinical Center of Vojvodina, Novi Sad
- Spain (2):
  - Hematologia Clínica, Barcelona
  - University Clinical Hospital of Salamanca, Department of Hematology, Salamanca